CLINICAL TRIAL: NCT04453228
Title: Analysis of the Mass Skiers' Injury in a Large Ski Resort in Chongli, China
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020108
Record Dates: First submitted 2020-06-25; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Skiing Injury
Keywords: Ski resorts; Skiing; Sports injury; The winter Olympics
MeSH Terms: conditions — Athletic Injuries | interventions — Statistics as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2017-2018 snow season: Injured skiers in the 2017-2018 snow season
  Interventions: Other: Classification statistics
- 2018-2019 snow season: Injured skiers in the 2018-2019 snow season
  Interventions: Other: Classification statistics

INTERVENTIONS:
Other: Classification statistics — We classified skiers in the two snow seasons by injury site, type of injury, cause of injury, etc

SUMMARY:
This study takes the injury situation of a large ski resort in Chongli during the 2017-2018 and 2018-2019 snow seasons as an example, aiming to preliminarily understand the injury situation of mass skiing in ski resorts in China, and provide a basis for predicting the rapidly growing medical demand for treatment and treatment of ski injuries in the context of 2022 Winter Olympic Games.

DETAILED DESCRIPTION:
Objective: To make a retrospective analysis of the injuries of skiing population in a large ski resort in Chongli, China and provide a basis for predicting the rapidly increasing medical needs for ski injuries in the context of the 2022 winter Olympic Games.

Methods: The basic data of all injured skiers who were treated in a medical station of a large ski resort in Chongli during the 2017-2018 and 2018-2019 snow seasons were collected. The number of skiers, the number of injuries, the causes of injuries, the types of injuries and the locations of injuries were compared.

ELIGIBILITY:
Inclusion Criteria:

* All of the injured in a snow season at a snow resort

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: During the 2017-2018 and 2018-2019 snow season, the injured skiers were amateurs.There were teenagers and teachers.But most of them were young and middle-aged.
Sampling Method: Non-Probability Sample
Enrollment: 753 (Actual)
Dates: Start 2020-03-22 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Injury rate during the snow season | Injury rate during a snow season,an average of 5 months
  This study statistically analyzed the injury rates of the two snow seasons to see if there was any difference

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No